CLINICAL TRIAL: NCT05576142
Title: Oral Findings in Pediatric Patients With Allergic Rhinitis and/or Asthma: a Cohort Study
Brief Title: Oral Findings in Pediatric Patients With Allergic Rhinitis and/or Asthma
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Other Study IDs: 2022-PEDORALFINDINGS
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Allergic Rhinitis; Asthma in Children; Dental Caries; Periodontal Diseases
MeSH Terms: conditions — Rhinitis, Allergic; Dental Caries; Periodontal Diseases | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Patients from this group were diagnosed from allergic rhinitis and/or asthma.
  Interventions: Diagnostic Test: Oral examination
- Control Group: Healthy children.
  Interventions: Diagnostic Test: Oral examination

INTERVENTIONS:
Diagnostic Test: Oral examination — Patients underwent oral examination with the recording of DMFT, PSR, PI and presence/absence of mouth breathing.

SUMMARY:
The aim of the study was to evaluate if there were differences in oral findings between patients diagnosed with allergic rhinitis and/or asthma and a control group of health people.

DETAILED DESCRIPTION:
The aim of the study was to evaluate if there were differences in oral findings between patients diagnosed with allergic rhinitis and/or asthma and a control group of health people. At the oral evaluation, the following indexes were calculated: PSR, Periodontal Screening and Recording; PI, Plaque Control Record and DMFT, Decayed Missing Filled Teeth Index. Absence or presence of mouth breathing was also recorded. Linear regressions were calculated to compare the oral findings with gravity of allergic rhinitis, to asthma compensation and to asthma treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 5-14 years old
* presence of allergic rhinitis diagnosed according to ASIA guidelines and/or presence of asthma diagnosed according to GINA guidelines

Exclusion Criteria:

* refuse to participate to the study
* presence of systemic diseases that could alter oral conditions (Sjögren syndrome, celiac disease, calcium disorders).

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients addressing to the Pediatric clinic of Fondazione IRCCS Policlinico San Matteo, Pavia, Italy for medical care.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
PSR - Periodontal Screening and Recording (Landry and Jean, 2002) | Baseline
  Scoring criteria:
  * 0: Absence of clinical signs
  * 1: Bleeding on probing
  * 2: Supra and/or subgingival calculus and/or defective margins
  * 3: Periodontal pocket 4 mm to 5.5 nm deep (coloured band on probe partially visible)
  * 4: Periodontal pocket 6 mm deep (colored band no longer visible)
  * *: Periodontal abnormalities present
  * X: Sextant absent or fewer than 2 teeth
PCR - Plaque Control Record (O' Leary et al., 1972) | Baseline
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.
DMFT - Decayed Missing Filled Teeth Index (WHO, 2013) | Baseline
  Sum of the decayed, missing, filled teeth.
Mouth breathing | Baseline
  Assessment of the presence/absence of mouth breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MSc, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data are available upon request to the Principal Investigator.